CLINICAL TRIAL: NCT04705948
Title: Comparing the Effect of Ketamine and Magnesium Sulfate Gargling With Placebo on Post-operative Sore Throat: A Randomized Controlled Trial
Brief Title: Comparing the Effect of Ketamine and Magnesium Sulfate Gargling With Placebo on Post-operative Sore Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Mechaal Benali, Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTEM POST
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Complications
Keywords: sore throat; Ketamine; magnesium sulfate; endotracheal intubation
MeSH Terms: conditions — Postoperative Complications; Pharyngitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine group (Experimental): ketamine gargle (0.5 mg/kg up to 30 ml dextrose water) 15 minutes before the operation
  Interventions: Drug: Magnesium sulfate versus ketamine
- magnesium sulfate group (Experimental): magnesium sulfate gargle (20 mg/kg up to 30 mL G5%) 15 minutes before the operation.
  Interventions: Drug: Magnesium sulfate versus ketamine

INTERVENTIONS:
Drug: Magnesium sulfate versus ketamine — Magnesium sulfate versus ketamine for of post-operative sore throat after endotracheal intubation
  Other Names: postoperative complication

SUMMARY:
A prospective randomized double-blind study including patients ASA I-II, aged more than 18 years undergoing surgery under general anesthesia (GA) and endotracheal intubation. Patients were randomized allocated into 2 groups: ketamine group received ketamine gargle (0.5 mg/kg up to 30 ml dextrose water) and magnesium group received magnesium sulfate gargle (20 mg/kg up to 30 mL dextrose water ) 15 minutes before the operation.

Our primary outcome is sore throat and the secondary judging criteria are cough, dysphonia and satisfaction. A standardized anesthesia protocol was followed for all patients. After extubation, the patients were asked to grade POST, hoarseness, and cough at 15 min, 1h, and 24 h.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized, double-blind study. the investigators included in the study the patients:

whose age is greater than or equal to 18 years; ASA class 1 or 2, proposed for elective visceral, orthopedic, oncology, ophthalmologic, urologic surgery under general anesthesia with orothracheal intubation, expected duration ≤ 120 min.

the non-inclusion criteria are known allergy to ketamine or maguisuim sulphate, ASA 3 and more, cervical surgery; rapid sequence induction, difficult intubation planned or history of difficult intubation, malformation of the O.R.L sphere; upper respiratory tract infections. the need for multiple laryngoscopies for orotracheal intubation (≥ 2 attempts); the need for a postoperative nasogastric tube.

randomization is performed upon entering the operating room. The gargle allocation scheme, Ketamine Group or Magnesium Sulfate Group was randomly generated using a randomization table with an allocation ratio of 1: 1.

Postoperative follow-up was carried out in the post-intervention monitoring room then in hospitalization within the various referring services (general surgery, orthopedics, O.R.L and ophthalmology).

On the day of the procedure, the doctor responsible for the study prepares the two types of solutions containing:

* One of magnesium sulfate (20mg / kg diluted in 30cc of 5% glucose serum);
* The other ketamine (50mg diluted in 30cc of 5% glucose serum). These two solutions were distributed over two groups of patients for use as a gargle, lasting at least 60 seconds for each patient in each group and 15 minutes before the surgery.

The primary endpoint is the incidence and severity of POST at the twenty-fourth hour postoperatively The secondary outcomes are the incidence and severity of POST at 15 minutes and one hour postoperatively; The occurrence of cough, The presence of dysphonia and Patient satisfaction

The severity of POST was scored on a three-point score from 0 to 2 (0 = No pain; 1 = Oropharyngeal pain on speaking; 2 = Spontaneous oropharyngeal pain)

ELIGIBILITY:
Inclusion Criteria:

* age is greater than or equal to 18 years
* ASA class 1 or 2
* patients proposed for elective visceral, orthopedic, oncology, ophthalmologic, urologic surgery under general anesthesia with orothracheal intubation

Exclusion Criteria:

* known allergy to ketamine or maguisuim sulphate
* ASA 3 and more
* cervical surgery
* difficult intubation planned or history of difficult intubation
* malformation of the O.R.L sphere
* the need for multiple laryngoscopies for orotracheal intubation (≥ 2 attempts);
* the need for a postoperative nasogastric tube.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-02-07 (Actual); Study Completion 2021-02-07 (Actual)

PRIMARY OUTCOMES:
severity of post-operative sore throat | at the twenty-fourth hour postoperatively
  The severity of POST was scored on a three-point score from 0 to 2 (0 = No pain; 1 = Oropharyngeal pain on speaking; 2 = Spontaneous oropharyngeal pain)

SECONDARY OUTCOMES:
Patient satisfaction | at the twenty-fourth hour postoperatively
  score of three points: satisfied (2 points); moderately satisfied (1 points); not satisfied (0 points)
the incidence of cough | at the twenty-fourth hour postoperatively
  no cough 0 point and presence 1 point

CONTACTS AND LOCATIONS:
Overall Officials: mechaal benali, PROFESSOR, Study Director — university manar Tunis tunisia
Locations (1):
- Mechaal Benali, Nabeul, Mrezga Hammamet, Tunisia

IPD SHARING:
Plan to Share IPD: No